CLINICAL TRIAL: NCT07248215
Title: The Effect of Newborn Basic Care Training Provided to Prospective Fathers Via a Website on Self-Efficacy and Perceptions of Spousal Support During Pregnancy
Acronym: ENBC-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Sevilay Ergun Arslanli, PhD, Lecturer, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CankırıKaratekinUniversity
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Social Support; Spouse; Self Efficacy; FATHER
Keywords: spousal; social support; newborn; father; self- efficacy

STUDY DESIGN:
Intervention Model Description: This research will be conducted as a prospective pretest-posttest, two-group (1:1), randomized controlled experimental design.In the study, expectant fathers and pregnant women will be assigned to experimental and control groups using the block randomization method. The block randomization process was conducted via the website https://www.randomizer.org/. Within the scope of block randomization, 35 separate blocks were initially created, with two individuals in each group. The assignment of individuals within the blocks to the case and control groups was based on random numbers generated by https://www.randomizer.org/. For example, in this table, the first couple who met the study inclusion criteria and volunteered to participate was assigned to the experimental group, the second couple to the control group, the third couple to the expert are blinded during data analysis and group assignment.
Who Masked: Participant, Outcomes Assessor
Masking Description: The researcher will not be informed of the group placement of expectant fathers and mothers according to the randomization table before data collection, and the researcher will be blinded during group assignment. The researcher, who will also provide the training, will be blinded during the assignment of fathers to groups, but will not be blinded during the training and evaluation phases. Once the data collection process is complete, the data will be transferred to a computer and analyzed by an expert independent of the research. This will ensure that the researcher and the independent expert are blinded during data analysis and group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Website (Experimental): In this study, a website called "https://www.bebeklerinbakimi.com/" was created, consisting of scale items developed using literature reviews, research results, evidence-based practice guidelines, and videos prepared in accordance with the booklet.
  Interventions: Behavioral: Web Group
- Routine Care (No Intervention): The researcher will not perform any neonatal care interventions in this group; they will continue to receive routine care at the midwifery school.

INTERVENTIONS:
Behavioral: Web Group — Fathers who agree to participate in the study will attend routine follow-up and training provided by the midwifery school during data collection, and then participate in baby care training provided by the researcher. These training sessions will be provided within the last three months of pregnancy for fathers whose wives are in their last trimester. This will allow the prospective fathers to learn how to use the website and log in for the first time under the researcher's guidance.
  Arms: Website

SUMMARY:
Support programs and training should be provided to parents by healthcare professionals, especially neonatal nurses and midwives, in line with these basic newborn care needs. Fathers, in particular, express a greater need for training because they feel less competent than mothers in newborn care. The concept of self-efficacy was first introduced by Bandura and defined as "individuals' beliefs in their capacity to organize and perform the actions necessary to perform assigned tasks". Self-efficacy is, in another definition, the belief that individuals have in themselves in the face of any situation they encounter, and these self-efficacy beliefs vary from situation to situation. If individuals have low self-efficacy, they will not find themselves competent in the situation they encounter and may not be able to do the task even if they have the capacity to do it. In this context, low self-efficacy levels of fathers in newborn care negatively affect their participation in care. During the prenatal period, expectant fathers' participation in childbirth preparation training and spending time with their partners allows them to focus on the baby and their partner's pregnancy. While the literature explores the emotions and experiences of pregnant women, studies on expectant fathers' cooperation during pregnancy, their self-efficacy for baby care, and their perception of spousal support are scarce. Therefore, this study aims to investigate the impact of basic newborn care training provided to expectant fathers with pregnant wives via a website on expectant fathers' self-efficacy and their wives' perception of spousal support during pregnancy.

DETAILED DESCRIPTION:
The neonatal period encompasses the first 28 days after birth. Babies born between 38 and 42 weeks are classified as term newborns, those born before 37 weeks as premature babies, and those born after 42 weeks as postmature babies. The newborn must experience physiological changes and adaptation in their body systems with birth. While completely dependent on the placenta for gas exchange, thermoregulation, nutrition, and excretion of metabolic products during the intrauterine period, they perform these functions independently after birth. However, because the newborn's systems are not fully developed like those of adults, they have difficulty performing these functions in the first days, and deviations from normal can occur within a short time. Therefore, ensuring and maintaining hemostasis in newborns is one of the primary goals of neonatal care. A baby's health and quality of care during the intrauterine, birth, and neonatal period affect their entire life. Therefore, a healthy newborn period, from birth to the intrauterine period, and optimally meeting their care needs will lay the foundation for the rest of their life. The most important of these care needs relate to the newborn's hygiene, safety, and nutrition. Support programs and training should be provided to parents by healthcare professionals, especially neonatal nurses and midwives, in line with these basic newborn care needs. Fathers, in particular, express a greater need for training because they feel less competent than mothers in newborn care. The concept of self-efficacy was first introduced by Bandura and defined as "individuals' beliefs in their capacity to organize and perform the actions necessary to perform assigned tasks". Self-efficacy is, in another definition, the belief that individuals have in themselves in the face of any situation they encounter, and these self-efficacy beliefs vary from situation to situation. If individuals have low self-efficacy, they will not find themselves competent in the situation they encounter and may not be able to do the task even if they have the capacity to do it. In this context, low self-efficacy levels of fathers in newborn care negatively affect their participation in care. Another study found that the self-efficacy levels of mothers and fathers in the intervention group improved after newborn care and parenting preparation training provided to parents in the early period through a mobile health application. Therefore, it is extremely important that fathers who care for newborns receive various trainings to increase their knowledge and skills about newborn care before and immediately after birth. During the prenatal period, expectant fathers' participation in childbirth preparation training and spending time with their partners allows them to focus on the baby and their partner's pregnancy. Furthermore, it has been reported that supporting their partners during pregnancy has a positive effect on the baby's cortisol levels in the intrauterine period and has a protective effect on the baby's health. It is emphasized that pregnant women often need spousal support during pregnancy and birth, that spousal support makes pregnancy less stressful, and that failure to provide adequate spousal support when needed can lead to irreversible problems. It has been reported that low perception of spousal support during pregnancy is associated with neonatal outcomes such as newborn weight, neonatal distress, and prematurity, and that it negatively affects mother-infant bonding and breastfeeding. While the literature explores the emotions and experiences of pregnant women, studies on expectant fathers' cooperation during pregnancy, their self-efficacy for baby care, and their perception of spousal support are scarce. Therefore, this study aims to investigate the impact of basic newborn care training provided to expectant fathers with pregnant wives via a website on expectant fathers' self-efficacy and their wives' perception of spousal support during pregnancy.

H11: Basic newborn care education provided to expectant fathers through the website has a positive effect on fathers' self-efficacy.

H21: Basic newborn care education provided to expectant fathers through the website has a positive effect on expectant mothers' perception of spousal support during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

The study required the following criteria for participating fathers:

* Their wife's pregnancy was in the third trimester
* They were over 18 and under 50
* They agreed to participate in the study and signed the voluntary consent form
* They had internet access on their phone
* They knew how to use a telephone
* They could read and understand Turkish
* They were oriented to place, time, and person
* They had no problems with their wife's pregnancy
* They had no communication or visual impairments.

The study included mothers who were:

Pregnant women were included if they:

* were over 18 but under 50 years old
* were in their third trimester of pregnancy
* agreed to participate in the study and signed the voluntary consent form
* knew how to use a telephone and had internet access on their phone
* could read and understand Turkish
* were oriented to place, time, and person
* had no communication or visual impairments.

Exclusion Criteria:

* participated in the study but did not wish to continue in the future
* had a child or spouse develop a health problem during the study period
* did not visit the website during their wife's pregnancy or did not follow the practices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-26 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | Before starting the study
  The Personal Information Form was developed by the researcher for both expectant fathers and expectant mothers by reviewing relevant literature. The form for expectant fathers consists of eight open-ended and closed-ended questions inquiring about fathers' socio-demographic and paternal characteristics. The form for expectant mothers consists of six open-ended and closed-ended questions inquiring about fathers' socio-demographic and paternal characteristics.
Fathers' Newborn Care Self-Efficacy Scale (BYBÖÖ) | The researcher administers the Fathers' Newborn Care Self-Efficacy Scale (FNSS) as a pre-test at the beginning of the study; the same scales are administered again at 3 months to collect post-test data.
  Ergün Arslanlı et al. (2024) developed the scale, which consists of three subscales (Hygiene, Safety, and Nutrition) and 17 items safety, and nutrition. The scale is a five-point Likert-type scale, with scores ranging from 17 to 85. Higher scores indicate higher father self-efficacy in basic newborn care.
Perception of Spousal Support During Pregnancy Scale (GEDAÖ) | The researcher administers the Fathers' Newborn Care Self-Efficacy Scale (FNSS) as a pre-test at the beginning of the study; the same scales are administered again at 3 months to collect post-test data.
  The scale consists of 16 items and three subscales. It can be used in studies with normal and high-risk pregnancies. The lowest possible score from the sixteen-item scale is 16, and the highest is 80. High scores on the scale should be interpreted as indicating high perceived spousal support during pregnancy, while low scores should be interpreted as indicating low perceived spousal support.

CONTACTS AND LOCATIONS:
Locations (1):
- ÇANKIRI KARATEKİN ÜNİVERSİTESİ SAĞLIK BİLİMLERİ FAKÜLTESİ Hemşirelik Bölümü, Çankırı, Çankırı Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shorey S, Ng YPM, Siew AL, Yoong J, Morelius E. Effectiveness of a Technology-Based Supportive Educational Parenting Program on Parental Outcomes in Singapore: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Jan 10;7(1):e4. doi: 10.2196/resprot.8062. PMID 29321127
- [Result] Shorey S, Dennis CL, Bridge S, Chong YS, Holroyd E, He HG. First-time fathers' postnatal experiences and support needs: A descriptive qualitative study. J Adv Nurs. 2017 Dec;73(12):2987-2996. doi: 10.1111/jan.13349. Epub 2017 Jun 21. PMID 28557020
- [Result] Ergun Arslanli S, Celebioglu A, Celik I, Uzun NB. Development and Psychometric Testing of the Fathers' Self-Efficacy Scale for Newborn Care. Asian Nurs Res (Korean Soc Nurs Sci). 2024 May;18(2):97-105. doi: 10.1016/j.anr.2024.04.001. Epub 2024 Apr 26. PMID 38677473